CLINICAL TRIAL: NCT06317766
Title: Histological Study of the Effects of a 2910 nm Fiber Laser Technology
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: FA Corporation (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UC 20-2023
Record Dates: First submitted 2024-01-30; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Skin Laxity
Keywords: Histology; 2910 nm Fiber Laser; Ablative Fractional Laser
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Part 1 Pre-Clinical Procedure (Experimental): * 1 healthy adult (male or female)
  * 18-75 years of age, who are scheduled to undergo an abdominoplasty (where abdominal skin will be excised) will be recruited.
  * Informed consent will be obtained by a delegated member of the study staff prior to the day of surgery.
  * On the day of the scheduled procedure, the laser device will be applied to the skin that will be removed as part of the surgery. The treatment will be completed after induction and prior to prepping for the surgical procedure.
  Interventions: Device: 2910 nm Fiber Laser Treatment; Pre-Clinical Histology Evaluation
- Part 2 Clinical Study Procedure (Experimental): * 1 healthy adult (male or female)
  * 18-75 years of age, who are scheduled to undergo an abdominoplasty (where abdominal skin will be excised) will be recruited.
  * Informed consent will be obtained by a delegated member of the study staff prior to the day of surgery.
  * The study team will utilize the specific setting based off the results of Part 1.
  * Subject will be asked to return to the site on days -30, -3, -2, -1 before their procedure.
  * At each visit, subjects will receive a single pulse treatment in areas that will be marked by the study team.
  * On the day of their procedure, a member of the study team will administer 1 final pulse immediately post-surgery and all 5 timepoints will be harvested for analysis.
  Interventions: Device: 2910 nm Fiber Laser Treatment; Part 2 Histology Evaluation

INTERVENTIONS:
Device: 2910 nm Fiber Laser Treatment; Pre-Clinical Histology Evaluation — Treatment with 2910 nm fiber laser focusing on its diverse energy settings and histological evaluation post abdominoplasty.
  Arms: Part 1 Pre-Clinical Procedure
Device: 2910 nm Fiber Laser Treatment; Part 2 Histology Evaluation — Healing Progression: Treatment with 2910 nm fiber laser focusing on its diverse energy settings and histological evaluation post abdominoplasty.
  Arms: Part 2 Clinical Study Procedure

SUMMARY:
The goal of this interventional clinical study is to conduct a comprehensive evaluation of the 2910 nm fiber laser focusing on its diverse energy settings. 2 subjects will be recruited for this 2 part histology study. The main This study will provide valuable insights into the device's capabilities and expand knowledge of its clinical utility. The first part of this study is intended to optimize treatment parameters based on observed effects at the molecular level. The second part will investigate the state of tissue at different timepoints following treatment.

Part 1 Pre-Clinical Study Procedure:

* 1 healthy adult (male or female)
* 18-75 years of age, who are scheduled to undergo an abdominoplasty (where abdominal skin will be excised) will be recruited.
* Informed consent will be obtained by a delegated member of the study staff prior to the day of surgery.
* On the day of the scheduled procedure, the laser device will be applied to the skin that will be removed as part of the surgery. The treatment will be completed after induction and prior to prepping for the surgical procedure.

Part 2 Clinical Study Procedure:

* 1 healthy adult (male or female)
* 18-75 years of age, who are scheduled to undergo an abdominoplasty (where abdominal skin will be excised) will be recruited.
* Informed consent will be obtained by a delegated member of the study staff prior to the day of surgery.
* The study team will utilize the specific setting based off the results of Part 1.
* Subject will be asked to return to the site on days -30, -3, -2, -1 before their procedure.
* At each visit, subjects will receive a single pulse treatment in areas that will be marked by the study team.
* On the day of their procedure, a member of the study team will administer 1 final pulse immediately post-surgery and all 5 timepoints will be harvested for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between 18-75 years of age.
* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements.
* Fitzpatrick skin types I-IV.
* Subjects who have pre-scheduled a body or facial contouring procedure.

Exclusion Criteria:

* Subjects with active localized or systemic infections
* Immunocompromised subjects
* Subjects with coagulation disorder
* History of radiation therapy to treatment area
* Subject with a history of lidocaine or ester-based local anesthetics
* Pacemaker or internal defibrillator
* Superficial or metal implants in the area
* Current or history of skin cancer, as well as any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders
* Pregnancy and nursing
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Diseases which may be stimulated by light at the wavelengths used, such as history of Systemic Lupus Erythematosus, Porphyria, and Epilepsy.
* Patients with a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regime.
* Any active condition in the treatment area, such as sores, psoriasis eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants.
* Use of medication and herbs known to induce photosensitivity to light exposure at the wavelengths used, such as Isotretinoin (Accutane) within the last 6 months, tetracyclines, or St. John's Wort within the last two weeks.
* Any surgical procedure in the treatment area within the last 3 months or before complete healing.
* Tattoo or permanent makeup in the treatment area.
* Excessively tanned skin from sun, tanning beds or tanning creams within last the two weeks.
* As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
TUNEL Staining | Up to 30 days
  Terminal deoxynucleotidyl transferase-mediated dUTP nick end labeling (TUNEL) is a robust technique for detecting apoptosis or cell death. Fluorescence intensity of the TUNEL positive cells in the treatment groups compare to control (untreated) will be measured. The data is given as fold change or percentage.
Mason's Trichrome | Up to 30 days
  The structural analysis using Trichrome will be observational to demonstrate any deviation from the normal skin structure (descriptive tool).

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Assa, President FACorp, Study Director — FA Corporation; Jeffrey Kenkel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Soutwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We are unsure of the current publication plan for this clinical study data. Due to IP and confidentiality we would like to request this filing remain private.